CLINICAL TRIAL: NCT03984461
Title: A Phase II, Randomized, Parallel-Group Study to Investigate the Combined Use of PRP with Lipoaspirate And/or Bone Marrow Aspirate in Osteoarthritis
Brief Title: The Combined Use of PRP with Lipoaspirate And/or Bone Marrow Aspirate in Osteoarthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Grant M. Pagdin (Other)
Responsible Party: Sponsor-Investigator, Dr. Grant M. Pagdin, Qualified Investigator, Pagdin Health
Organization: Pagdin Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OASC2015
Record Dates: First submitted 2019-05-28; First posted 2019-06-13 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Platelet Rich Plasma (PRP); Micronized Lipoaspirate (MAT); Bone Marrow Aspirate (BMA)
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Group A - PRP plus Lipoaspirate Group B - PRP plus Bone Marrow Aspirate Group C - PRP plus Lipoaspirate plus Bone Marrow Aspirate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A - PRP plus Lipoaspirate (Active Comparator): Equal proportions of PRP plus micronized adipose tissue (lipoaspirate). Total Volume varies by joint.
  Interventions: Biological: Autologous cell therapy
- Group B - PRP plus Bone Marrow Aspirate (Active Comparator): Equal proportions of PRP plus bone marrow aspirate. Total Volume varies by joint.
  Interventions: Biological: Autologous cell therapy
- Group C - PRP plus Lipoaspirate plus Bone Marrow Aspirate (Active Comparator): Equal proportions of PRP plus micronized adipose tissue (lipoaspirate) plus bone marrow aspirate. Total Volume varies by joint.
  Interventions: Biological: Autologous cell therapy

INTERVENTIONS:
Biological: Autologous cell therapy — Biologic material is harvested from the participant and re-injected into an osteoarthritic joint

SUMMARY:
To demonstrate the efficacy of the combined use of platelet-rich plasma (PRP) with lipoaspirate and/or bone marrow aspirate in osteoarthritis of major joints, and to compare the outcomes achieved using three combinations: PRP plus lipoaspirate, PRP plus bone marrow aspirate, and PRP plus both lipoaspirate and bone marrow aspirate.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the efficacy of the combined use of platelet-rich plasma (PRP) with lipoaspirate and/or bone marrow aspirate in osteoarthritis of major joints, and to compare the outcomes achieved using three combinations: PRP plus lipoaspirate, PRP plus bone marrow aspirate, and PRP plus both lipoaspirate and bone marrow aspirate.

A total of 240 participants will be randomly assigned to one of three treatment groups: Group A will receive PRP plus lipoaspirate, Group B will receive PRP plus bone marrow aspirate, and Group C will receive tri-partite therapy of PRP + lipoaspirate + bone marrow aspirate which allows for 80 in each group. The combination of biologic materials will be injected in to an arthritic joint.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing written informed consent and willing and able to adhere to all protocol requirements.
2. Male or female at least 19 years of age at the time of providing written informed consent.
3. Evidence of OsteoArthritis in a major joint requires recent (within one year) imaging, either by x-ray or MRI. Kellgren & Lawrence Grades 1-3 are accepted for participation.

Exclusion Criteria:

1. BMI > 35
2. Arthroscopic surgery to the treatment joint within 12 months
3. Cortisone or HA injection within the last 3 months prior to stem cell injection
4. Inability to hold antiplatelet therapy according to treating provider prior to procedure
5. Kellgren & Lawrence Grade 4 Osteoarthritis
6. Participants with a platelet count less than 100 x 109
7. Participants with a Hemoglobin less than 100 g/L
8. Participants who have an active Infection with fever and/or elevated white blood cell (WBC) count
9. Participants with an active Cancer diagnosis.
10. Participants with autoimmune disorders including rheumatoid arthritis and lupus.
11. Women who are pregnant will be excluded due to the possibility of fetal harm associated with x-rays. Should a participant become pregnant during the study, she will be withdrawn from further treatment and imaging, but can participate in symptom follow-up. Female participants of childbearing potential will be counseled at screening about contraception and encouraged to use birth control for the duration of the study.
12. Participants with allergies to lidocaine, heparin, or epinephrine.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline through to end of study for the Visual Analogue Scale (VAS). | The VAS will be measured at baseline (week 1) through to the end of the study (week 104). To test for improvement, comparisons to baseline will be made at 6 months (week 26,) 12 months (week 52) and 24 months (week 104).
  Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity. This scale measures ranges from 0 whereby the patient has no discomfort or distress to 10 where the patient has agonizing pain and is in unbearable distress. (0 - None, 1, 2 - Annoying, 3, 4 - Uncomfortable, 5, 6 - Dreadful, 7, 8 - Horrible, 9, 10 - Agonizing). The patient can place an x anywhere on the continuum between 0-10 based on their level of discomfort . We will then measure the scale using a ruler to the tenth of a point. The VAS scale will be completed at each visits 2-7. Comparisons will be made from baseline to end of study to determine the overall improvement.
Changes from baseline through to the end of study for the Short Form 12 item version 2 (SF12-v2) | The SF12-v2 will be measured at baseline (week 1) through to the end of the study (week 104). To test for improvement, comparisons to baseline will be made at 6 months (week 26,) 12 months (week 52) and 24 months (week 104).
  The SF-12 is a validated and widely used twelve question health survey used to assess health related quality of life from the patients perspective. The SF12-v2 items are scored so that a higher score means a better health. For example, the functioning items are scored so that a higher score represents better functioning, whereby pain items scored so that a high score indicates freedom from pain. The SF12-v2 will be completed at each visits 2-7. Comparisons will be made from baseline to end of study to determine the overall improvement.

SECONDARY OUTCOMES:
Comparison to evaluate the degree of change among treatment arms (Group A, Group B and Group C) from baseline visit through to end of study. | The VAS will be measured at baseline (week 1) through to the end of the study (week 104). To test for improvement, comparisons to baseline will be made at 6 months (week 26,) 12 months (week 52) and 24 months (week 104).
  To evaluate the variations among the three treatment arms (lipoapirate [group A], bone marrow aspirate [group B], and lipoasiprate and bone marrow aspirate [group c] we will use the overall average of the VAS for each group. It is the investigator's hypothesis that we anticipate that group c might have a superior outcome to either group A or group B.
Comparison to evaluate the degree of change among treatment arms (Group A, Group B and Group C) baseline visit through to end of study. | The SF12-v2 will be measured at baseline (week 1) through to the end of the study (week 104). To test for improvement, comparisons to baseline will be made at 6 months (week 26,) 12 months (week 52) and 24 months (week 104).
  To evaluate the variations among the three treatment arms (lipoapirate [group A], bone marrow aspirate [group B], and lipoasiprate and bone marrow aspirate [group c] we will use the overall average of the SF12-v2 for each group. It is our hypothesis that we anticipate that group c might have a superior outcome to either group A or group B.
Flow cytometry | Visit 2 (Week 1) Samples are collected at visit 2 (week 1) and sent away for analysis by a university. The results will be received from the university prior to end for overall data analysis.
  Numbers and viability of stem cells

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Rosenfeld, MD, Study Chair — Quorum Review IRB
Locations (1):
- Pagdin Health, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No